CLINICAL TRIAL: NCT05824780
Title: Functional and Performance Effects of a 4-week Weightlifting Program in Highly Trained Adolescent Basketball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Universidad Europea de Valencia (Other)
Responsible Party: Principal Investigator, Fernando Domínguez-Navarro, Clinical Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-1523453
Record Dates: First submitted 2023-02-08; First posted 2023-04-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Athletic Injuries
Keywords: Weighlifting; Strength; Functional outcomes; Adolescent; Basketball
MeSH Terms: conditions — Athletic Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two arms
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded to participants group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weigthlifting (Experimental): It consists of a 4-week strength training program based on weightlifting. Participants received previously education-training program on how to correctly perform the technique.
  Interventions: Other: Exercise training
- Plyometric training (Active Comparator): It consists of a 4-week strength training program based on plyometric exercises.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — 4-week weightlifting strength training

SUMMARY:
Weightlifting is an increasingly used intervention in the sport field to improve both function and performance outcomes. However, the effects in a pediatric and adolescent population are not well described, and require further research to elucidate the benefits and potential adverse effects compared to other strength training methods, such as plyometric training.

DETAILED DESCRIPTION:
Highly trained male and female adolescent basketball athletes aged 12-16 years will be recruited for the study. Participants will be randomly assigned to a 4-week program (12 sessions) of weightlifting or plyometric training. The training programs will be identical in sets and repetitions, progressively evolving each week towards fewer sets and fewer repetitions. The training intensity will be the same in both groups, calculated from the RM, starting at 70% in the first week and progressing by 5% each week until a final intensity of 85% in the last week. Therefore, both interventions evolve towards sessions with fewer sets and repetitions and higher loads.

The weightlifting intervention refers to the performance of highly technical and explosive multi-joint strength exercises. The program consists of six basic weightlifting maneuvers (hang power clean, overhead squat, hang power snatch, clean, split jerk, snatch), two of which are performed in each of the three weekly sessions. The order of execution of the exercises in the weekly sessions is always the same. To ensure the correct execution of the maneuvers, before starting the intervention, a brief familiarization program will be carried out. This consists of an explanation of the exercises by the research staff and practice by the participants with simultaneous correction.

The plyometric program follows the same structure, consisting in a total of 6 exercises (Max countermovement jump, double leg side jump, maximum squat jump, dropjump (20cm), single leg hurdle jump, doble leg multi hop) performed in groups of 2 for each weekly training session.

The design of the intervention program is based on previously published related articles.Training sessions will be supervised by a member of the research team with expertise in strength and conditioning in basketball athletes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy highly-trained basketball athletes

Exclusion Criteria:

* Current injury or complaining limiting sports activity
* No histoy of injury receiving non-operative treatment in the last 3 months
* No history of injury receiving operative treatment in the last 9 months
* Subjects who have previously carried out weightlifting training for at least 4 weeks of duration.
* Subjects physically unable to perform a strength training program

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline Repetition Maximum at 5 weeks | (I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  It refeers to the maximum weight that an athlete can lift correctly in one repetition. The maximum weight lifted is recorded in kg.
Change from baseline Hand Grip at 5 weeks | (I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  Measured with validated dynamometer equipment, it register the isometric strength that an athlethe perform in a hand grip contraction. Strength is recorded in kg. Three valid measures will be recorded and the mean value will be calculated.
Change from baseline Lower-limb muscle strength at 5 weeks | I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  Force Frame system equipment will be used to assess the isometric strength for lower-limb (hip and knee) muscles. Strength values will be expressed in kg. Three valid measures will be recorded and the mean value will be calculated.

SECONDARY OUTCOMES:
Change from baseline Ankle Mobility at 5 weeks | (I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  Check-your motion (R) device (validated) will be used to evaluate ankle dorsiflexion in weigth-bearing. position.Three valid measures will be recorded and the mean value will be calculated. Results will be expressed in cm
Change from baseline 20 meters Sprint at 5 weeks | (I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  From motion cameras, the time (seconds) that an athlete takes to perform a straight line movement of 20 meters at maximum speed will be recorded.
Change from baseline Counter movement jump (CMJ) test at 5 weeks | (I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  CMJ will be used as perfomance-based outcome. Athlete, in standing position, will perform a maximum vertical jump with both hands placed on the hips. The data will be collected with the Chronojump contact platform equipment, (Boscosystem®, Barcelona, Spain), registering the flight height (cm) and power (watts). Three valid measures will be recorded and the mean value will be calculated.
Change from baseline Hop test distance at 5 weeks | (I) Baseline: previous week before starting intervention, and (II) 5 weeks after baseline
  This test will be used to evaluate longitudinal maximum hop performance, registering the distance reached in cm. The procedure will be performed unilaterally with both legs. A tape measure will be used to record the distance traveled. Three valid measures will be registered and the mean will be calculated
Weight | Baseline
  Weight will be recorded from a validated electronic scale, expressed in kg.
Height | Baseline
  The height of the athletes will be measured using the vertical tape measure of a manual scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Domínguez Navarro, Valencia, Spain